CLINICAL TRIAL: NCT00048282
Title: HIV Prevention Preparedness Study
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Other Study IDs: HIVNET/HPTN 055
Record Dates: First submitted 2002-10-29; First posted 2002-10-30 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2006-01

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Incidence; HIV Seroprevalence; Vagina; Anti-Infective Agents; Administration, Topical; Gels; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to provide researchers with information that will help them prepare for a future study to test the efficacy of two anti-HIV vaginal gels. This study will also estimate how likely people living in certain areas are to become infected with HIV and other infections passed during sex.

DETAILED DESCRIPTION:
This study is designed to prepare for the implementation of a second study, HPTN 035: A Phase II/III Safety and Effectiveness Study of the Vaginal Microbicides BufferGel and PRO 2000/5 Gel (P) for the Prevention of HIV Infection in Women. HPTN 035 requires an average HIV seroincidence rate of 5-6 percent among enrolled participants. The primary objective of the present study is to estimate the rates of HIV seroincidence among women targeted for inclusion in HPTN 035.

Women will be enrolled in this study for 6 to 12 months. Study visits will take place monthly. At each visit, participants will complete a medical/menstrual history and undergo pregnancy testing. Each quarter, participants will undergo a structured interview about sexual practices and will receive HIV and STD tests, education, and counseling. Participants will also undergo a pelvic exam with wet mount testing for bacterial vaginosis, candidiasis, and trichomoniasis. Colposcopic evaluations will be performed at selected sites. Pap smears will be performed at sites with the capacity and expertise to prepare and interpret the smears and provide appropriate follow-up care to participants with abnormal results.

ELIGIBILITY:
Inclusion criteria:

* Sexually active (defined as having had vaginal intercourse at least once in the 3 months prior to screening).
* HIV-uninfected at screening.
* Able and willing to provide adequate locator information for study retention purposes.

Exclusion criteria:

* History of adverse reaction to latex.
* Non-therapeutic injection drug use in the 12 months prior to screening.
* Vaginal intercourse more than an average of 2 times per day in the 2 weeks prior to screening.
* Plans to travel away from the study site for more than 3 consecutive months in the next 12 months.
* Plans to relocate away from the study site in the next 12 months.
* Pregnancy or plans to become pregnant in the next 12 months.
* Pregnancy within 42 days prior to enrollment.
* Enrollment in any other study of a vaginally-applied product.
* Clinically apparent pelvic exam finding involving deep epithelial disruption.
* Diagnosis with a current STD and/or other reproductive tract infection requiring treatment.
* Conditions that would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200

CONTACTS AND LOCATIONS:
Overall Officials: Saidi Kapiga, MD, MPH, SCD, Study Chair — Harvard School of Public Health (HSPH); Gita Ramjee, PhD, Study Chair — South Africa Medical Research Council; Stephen Weiss, PhD, Study Chair — University of Miami
Locations (10):
- South Africa (4):
  - R.K. Khan Hospital, Chatsworth
  - Durban
  - Medical Research Council, Hlabisa
  - Hlabisa
- Tanzania (2):
  - Kilimanjaro Christian Med Ctr, Moshi
  - Moshi
- Zambia (4):
  - Chililabombwe
  - Chilenje Clinic, Lusaka, Sambia, Lusaka
  - Kamwala Clinic, Lusaka
  - Lusaka

REFERENCES:
- [Result] Kapiga S, Kelly C, Weiss S, Daley T, Peterson L, Leburg C, Ramjee G. Risk factors for incidence of sexually transmitted infections among women in South Africa, Tanzania, and Zambia: results from HPTN 055 study. Sex Transm Dis. 2009 Apr;36(4):199-206. doi: 10.1097/OLQ.0b013e318191ba01. PMID 19265734
- [Result] Ramjee G, Kapiga S, Weiss S, Peterson L, Leburg C, Kelly C, Masse B; HPTN 055 Study Team. The value of site preparedness studies for future implementation of phase 2/IIb/III HIV prevention trials: experience from the HPTN 055 study. J Acquir Immune Defic Syndr. 2008 Jan 1;47(1):93-100. doi: 10.1097/QAI.0b013e31815c71f7. PMID 17984760
- [Result] Schreiber CA, Sammel M, Hillier SL, Barnhart KT. A little bit pregnant: modeling how the accurate detection of pregnancy can improve HIV prevention trials. Am J Epidemiol. 2009 Feb 15;169(4):515-21. doi: 10.1093/aje/kwn345. Epub 2008 Dec 18. PMID 19095756